CLINICAL TRIAL: NCT00689715
Title: Long Term Outcomes After EUS-guided Ablation for Cystic Tumors of the Pancreas
Acronym: EUS-EP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dong Wan Seo, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0183
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Tumors of the Pancreas
Keywords: Cystic tumor; Pancreas; EUS
MeSH Terms: conditions — Neoplasms, Cystic, Mucinous, and Serous | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EP (Experimental): Single treatment arm
  Interventions: Procedure: Endoscopic ultrasonography-guided ethanol lavage with paclitaxel injection

INTERVENTIONS:
Procedure: Endoscopic ultrasonography-guided ethanol lavage with paclitaxel injection — A curvilinear-array echoendoscope and a 22 gauge needle were then used for cyst fluid aspiration, ethanol lavage and paclitaxel injection. The maximum possible volume of cyst fluid was aspirated, and the needle tip was carefully maintained inside the cyst to avoid parenchymal injury. Ethanol was injected into the collapsed cyst until the original shape was restored, and a lavage was then performed for 3-5 minutes. Pure ethanol (99%) was used for all patients except the first 2 in whom 88% ethanol was used. After reaspiration of the injected ethanol, the cyst cavity was injected with a solution containing 3 mg/mL paclitaxel and the needle then carefully retracted. The high viscosity of paclitaxel necessitated dilution in 0.9% normal saline for administration via a 22G needle. The volume of the paclitaxel solution administered was the same as the volume of the cyst fluid aspirated.
  Other Names: paclitaxel (Taxol®, 6 mg/mL, Bristol-Myers Squibb Pharmaceutical Group)

SUMMARY:
Cystic lesions of the pancreas are defined as round, fluid-filled structures within the pancreas detected by radiologic imaging. With widespread use of cross-sectional imaging modalities for various indications, such lesions are now detected in nearly 20% of abdominal imagings, with the majority discovered incidentally. These lesions encompass a wide spectrum of histopathologic entities and biologic behavior, ranging from benign to malignant. Substantial morphologic overlap restricts the accuracy in diagnosing specific type of cystic lesion in spite of recent advances in diagnostic modalities. It is a challenging issue to differentiate each cystic lesion and make a management plan since cystic lesions that are relatively common and asymptomatic may possess malignant potential. Although inflammatory pseudocysts were thought to account for 80-90% of cystic lesions of the pancreas, with cystic tumors accounting for the remaining,10 the latter may occur much more frequently than traditionally estimated.

To date, surgical resection is generally recommended for malignant and potentially malignant lesions. However, surgical resection of the pancreas still carries substantial morbidity and sometimes mortality, especially for the cystic lesion located in the head portion. Therefore, management should be individualized by risk-benefit analysis for each patient.

Recently, a pilot study of EUS-guided ethanol lavage for cystic tumors of the pancreas reported that complete resolution was achieved in only one-third of patients even though epithelial lining ablation was demonstrated in all resected specimens. Therefore, more effective treatment modalities or ablation agents are required to improve treatment responses. Intratumoral or intraperitoneal injection of chemotherapeutic agent has been used for endobronchial lesions of lung cancer, brain tumors and advanced ovarian cancer.13-16 EUS-guided injection of antitumor material has been reported in advanced pancreatic cancer. Although local injection of chemotherapeutic agents into pancreatic cystic tumors has not yet been reported, it is reasonable to suggest that such an approach may have an additive effect on ablation of the epithelial lining of cystic tumor when combined with ethanol lavage.

Paclitaxel, a widely used chemotherapeutic agent, inhibits cell processes that are dependent on microtubule turnover. Due to its highly hydrophobic nature,19 paclitaxel is expected to exert its effect longer when instilled within a closed cavity such as a cyst. The hydrophobic and viscous nature of paclitaxel may reduce the possibility of it leaking through a puncture site and causing complications.

The present study evaluated safety, feasibility and response following EUS-guided ethanol lavage with paclitaxel injection (EUS-EP) for treating cystic tumors of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* uni- or oligo-locular cystic tumors
* indeterminate cystic tumors for which EUS-guided fine needle aspiration (FNA) was required to obtain additional information
* cystic tumors that increased in size during the observation period

Exclusion Criteria:

* cystic tumors which had the typical morphology of serous cystadenomas (i.e., honeycomb appearance) and pseudocysts (i.e., parenchymal changes)
* evidence of communication between the cystic lesion and the main pancreatic duct according to endoscopic retrograde pancreatograms
* overt carcinomas with peripancreatic invasion
* patients with a bleeding tendency (prothrombin time > 1.5 international normalized ratio [INR] or platelet count < 50,000/μL).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events Treatment response by change of calculated cyst volume | early (< 7 days) and late (> 7days) adverse events
recurrence during follow up | any recurrence of cyst after complete resolution during at least 3 years follow up

SECONDARY OUTCOMES:
treatment response | 1 year
predictive factors for complete resolution | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wan Seo, M.D., Ph.D, Principal Investigator — Asan Medical Center, University of Ulsan Collge of Medicine
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Oh HC, Seo DW, Lee TY, Kim JY, Lee SS, Lee SK, Kim MH. New treatment for cystic tumors of the pancreas: EUS-guided ethanol lavage with paclitaxel injection. Gastrointest Endosc. 2008 Apr;67(4):636-42. doi: 10.1016/j.gie.2007.09.038. Epub 2008 Feb 11. PMID 18262182